CLINICAL TRIAL: NCT04965740
Title: EMPOWER Study: Exploring Medically Perceived Benefits, Use and Interest in Psychedelics and Cannabinoids: Observational Study With First Responders and Military Personnel Examining Previous Use Experience and Interest in Participating in Future Research Studies
Brief Title: Exploring Medically Perceived Benefits, Use and Interest in Psychedelics and Cannabinoids
Acronym: EMPOWER
Status: Completed | Type: Observational
Sponsor: Empower Research Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EMP-SURVEY-001
Record Dates: First submitted 2021-07-04; First posted 2021-07-16 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: PTSD; Anxiety; Anxiety Disorders; Depression; Depressive Disorder; Psychological; Psychedelic Experiences; Psychedelic Drug Dependence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Depressive Disorder | interventions — nabiximols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- North American First Responders: Spread directly to union representatives for email and messaging to those interested in taking the survey
  Interventions: Drug: Cannabis
- Oceana and European first responders: First responder unions and groups that are located outside of North America - particularly Australia, New Zealand, United Kingdom, other commonwealth nations.
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Recreational Cannabis
  Other Names: Recreational Cannabis

SUMMARY:
The primary objective of this study is to collect insights from first responders and military personnel on their need for, use of, and interest in physical and/or mental health medical marijuana or psychedelic-assisted therapy programs. These preliminary data will help to inform and guide the development of a larger patient-oriented study and the design of a clinical program geared towards enhancing therapy treatments for first responders and military personnel.

DETAILED DESCRIPTION:
Members of first response teams including police, firefighters, paramedics, and military personnel in Canada, the United States, Oceana, and Europe will be asked to participate. The majority of these teams are unionized, consisting of municipal, provincial and federally organized unions throughout Canada, United States, Oceana and Europe.

Whenever possible, the research team will provide an invitation to its members via union representatives. These unions are a trusted source for first responders and military personnel as they are intended to have the best interests of these first responders in mind. The union representatives possess the contact information of the first responders and military personnel. The unions routinely circulate e-mails to members that include information relevant for members such as upcoming events, important meetings, team activities on and off-duty, and opportunities to participate in research.

Emails with the link to the survey will be circulated to members approximately every month for 3 months, or until at least 1000 participants have responded. The link to the survey may also be shared through personal connections among first responders and/or word of mouth.

Participants will be sent a link to open an anonymous survey which they can complete at their location and time of choosing. Once the survey link has been accessed by a potential participant, background information will be provided regarding the project that includes an informed consent statement. Participants may leave the survey at any time should they wish to discontinue.

The survey will be distributed to first responders and military personnel using an online questionnaire. This survey will contain questions about basic demographics, history of mental health conditions, satisfaction with current life status, past use of cannabis and other psychedelic substances, and interest and potential barriers in trying psychedelic or medical marijuana-assisted physical or mental health therapy in a research or clinical context. The Brief Inventory of Psychosocial Functioning (13) and a subset of questions from the National Institute on Drug Abuse (NIDA) Quick Screen (14) have been integrated into the survey to enhance reliability and validity of results.

The survey will take approximately 15 minutes to complete. Once the survey has been submitted, participants will have the option to click a link to enter their email address using a separate collection form, if they would like to be contacted for future research opportunities.

The list of email addresses will not be linked to the survey results.

Data will be analyzed from all completed (fully or partially) and submitted surveys. Every question will contain a "Prefer Not to Say" option if a response is mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Adult (19+) first responders and military personnel in Canada, USA, Oceana and Europe -
* Not restricted by restricted by sex, gender, or diagnoses.
* Respondents must be able to read and write in English to participate.

Exclusion Criteria:

* Individuals who are not first responders, military personnel, or an aligned profession
* Individuals under the age of 19
* Those who are not able to read and write in English

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 10,000 first responders and/or military personnel will be asked to participate in the survey.
  Assuming a 20-30% response rate, the investigators expect approximately 2500 individual responses.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Collect Insights from First Responders | 8 months
  The primary objective of this study is to collect insights from first responders and military personnel on their need for, use of, and interest in physical and/or mental health medical marijuana or psychedelic-assisted therapy programs. These preliminary data will help to inform and guide the development of a larger patient-oriented study and the design of a clinical program geared towards enhancing therapy treatments for first responders and military personnel.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Potentially available for use in planning research with these groups

REFERENCES:
- [Background] Brunello N, Davidson JR, Deahl M, Kessler RC, Mendlewicz J, Racagni G, Shalev AY, Zohar J. Posttraumatic stress disorder: diagnosis and epidemiology, comorbidity and social consequences, biology and treatment. Neuropsychobiology. 2001;43(3):150-62. doi: 10.1159/000054884. PMID 11287794
- [Background] Marmar CR, McCaslin SE, Metzler TJ, Best S, Weiss DS, Fagan J, Liberman A, Pole N, Otte C, Yehuda R, Mohr D, Neylan T. Predictors of posttraumatic stress in police and other first responders. Ann N Y Acad Sci. 2006 Jul;1071:1-18. doi: 10.1196/annals.1364.001. PMID 16891557
- [Background] Jerome L, Feduccia AA, Wang JB, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Long-term follow-up outcomes of MDMA-assisted psychotherapy for treatment of PTSD: a longitudinal pooled analysis of six phase 2 trials. Psychopharmacology (Berl). 2020 Aug;237(8):2485-2497. doi: 10.1007/s00213-020-05548-2. Epub 2020 Jun 4. PMID 32500209
- [Background] Passie T, Emrich HM, Karst M, Brandt SD, Halpern JH. Mitigation of post-traumatic stress symptoms by Cannabis resin: a review of the clinical and neurobiological evidence. Drug Test Anal. 2012 Jul-Aug;4(7-8):649-59. doi: 10.1002/dta.1377. Epub 2012 Jun 26. PMID 22736575
- [Background] Gasser P, Holstein D, Michel Y, Doblin R, Yazar-Klosinski B, Passie T, Brenneisen R. Safety and efficacy of lysergic acid diethylamide-assisted psychotherapy for anxiety associated with life-threatening diseases. J Nerv Ment Dis. 2014 Jul;202(7):513-20. doi: 10.1097/NMD.0000000000000113. PMID 24594678
- See also: Survey Link — https://www.surveymonkey.com/r/empower-research-survey